CLINICAL TRIAL: NCT02840019
Title: Advanced Fetal Imaging - Phase II
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Massachusetts Institute of Technology (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Ellen Grant, Professor, Boston Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: R01EB017337 (NIH)
Record Dates: First submitted 2016-07-13; First posted 2016-07-21 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy
Keywords: Fetal MRI; Pregnancy; Pregnant Women; MRI Coil; MRI Sequence Development/Testing; Abnormal Fetuses; Typically Developing Fetuses; Fetal MRI Technology Development
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 60 minute research full MRI scan (Experimental): Pregnant women who are able to have an MRI are eligible for the 60 minute research full MRI scan. Pregnant women may have a healthy pregnancy, a concern for fetal/placental abnormalities with a clinical fetal MRI ordered by their doctor, or a concern for fetal/placental abnormalities without a clinical fetal MRI ordered by their doctor.
  The investigational MRI coil designed for pregnant women and research MRI sequences will be tested during the 60 minute research scan.
  Interventions: Device: Investigational MRI coil designed for pregnant women; Procedure: MRI Scan
- 15 minute research add-on MRI scan (Experimental): Pregnant women with a concern for fetal/placental abnormalities with a clinical fetal MRI at Boston Children's Hospital are eligible for the 15 minute research add-on MRI scan.
  The research MRI sequences will also be tested during the add-on research MRI scan.
  Interventions: Procedure: MRI Scan

INTERVENTIONS:
Device: Investigational MRI coil designed for pregnant women — The investigational MRI receiver coil designed specifically for pregnant women will be used during the 60 minute full research MRI scan. An MRI receiver coil is part of the MRI machine that is placed over the body part being imaged during every MRI scan. A coil is required to obtain MR images, yet there isn't one designed for pregnant women. This investigational MRI receiver coil for pregnant women will be tested to see if it helps improve image quality and take images faster.
  Arms: 60 minute research full MRI scan
Procedure: MRI Scan — All participants will participate in an MRI scan. The add-on MRI scan will be 15 minutes. The full MRI scan will be 60 minutes.

SUMMARY:
The goal of Advanced Fetal Imaging - Phase II is to advance fetal MRI imaging by designing MRI coils specifically for pregnant women and testing recently developed MRI image acquisition techniques. The investigators aim to more reliably obtain higher quality fetal MRI images when compared to current clinical fetal MRI.

DETAILED DESCRIPTION:
The main aim of this project is to evaluate and optimize the existing clinical magnetic resonance (MR) techniques for fetal imaging, and to also implement and test new MR technologies that would improve fetal imaging in general. This involves the development of new pulse sequences and image acquisition schemes that "freeze" fetal motion and hence provide improved image quality and robustness for both structural (T1- and T2- weighted, susceptibility and FLAIR imaging) and physiological imaging (diffusion, perfusion, spectroscopy, resting-state functional MRI, etc). The scope of this project also includes testing of newly developed radio frequency (RF) receive-only coil arrays that would inherently provide the means for faster imaging of the fetus, and thus complement the software developments.

ELIGIBILITY:
Inclusion Criteria:

* 60 Minute Full Research MRI Scan:

  * Gestational age between 18 and 40 weeks

    * AND
  * Pregnant women with a healthy pregnancy

    * OR
  * Pregnant women with a concern for fetal/placental abnormalities referred for a clinical fetal MRI by their obstetrician

    * OR
  * Pregnant women with a concern for fetal/placental abnormalities NOT referred for a clinical fetal MRI by their obstetrician
* 15 Minute Add-On Research Scan:

  * Gestational age between 18 and 40 weeks

    * AND
  * Pregnant women with a concern for fetal abnormalities referred for a clinical fetal MRI by their obstetrician

    * AND
  * The clinical fetal MRI will occur at Boston Children's Hospital

Exclusion Criteria:

* Pregnant women with a contraindication to MRI (implanted metal, non-removable piercings, pacemaker, etc)
* Pregnant women who are claustrophobic
* Pregnant women who are medically unstable for an MRI

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-07; Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Research fetal MRI image quality compared to standard clinical fetal MRI image quality | July 2016-December 2019, up to 41 months
  Research fetal MRI image quality will be compared to the standard clinical fetal MRI image quality.

SECONDARY OUTCOMES:
Research fetal MRI image quality compared to standard obstetric ultrasound image quality | July 2016-December 2019, up to 41 months
  Research fetal MRI image quality will be compared against standard obstetric ultrasound image quality.
Research MRI physiological data compared against standard obstetric physiological data obtained from ultrasound | July 2016-December 2019, up to 41 months
  Research fetal MRI physiology data (flow, perfusion, oxygen consumption) will be compared against standard obstetric physiological data obtained from ultrasound (e.g. Doppler measures).

CONTACTS AND LOCATIONS:
Overall Officials: P. Ellen Grant, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No